CLINICAL TRIAL: NCT06459375
Title: Comparative Effects of Modified Otago Exercises and Action Observation Training on Strength, Functional Mobility and Fall Risk in Patients With Diabetic Neuropathy
Brief Title: Effects of Modified Otago Versus Action Observation on Strength, Mobility and Fall Risk in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0283
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Neuropathies; Mobility; Fall
Keywords: Diabetic Neuropathies; Mobility; Fall
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: after randomization patients will be divided into two groups through computer generated number programme. Patients in group A will receive modified Otago exercises with conventional treatment. Patients in group B will receive Action Observation Training with conventional treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Otago exercise group (Experimental): patients in this group will receive modified Otago exercises with conventional treatment.
  Interventions: Other: modified otago exercises
- Action Observation Training group (Active Comparator): patients in this group will receive Action Observation Training with conventional treatment.
  Interventions: Other: Action Observation Training

INTERVENTIONS:
Other: modified otago exercises — patients will receive modified Otago exercises with conventional treatment.
  Arms: Modified Otago exercise group
Other: Action Observation Training — Patients will receive Action Observation Training with conventional treatment.
  Arms: Action Observation Training group

SUMMARY:
To compare the Effects of Modified Otago Exercise and Action Observation Training on strength, functional mobility and fall risk in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial. A total of 38 participants with diabetic neuropathy will be taken. By using non probability convenience sampling technique patients will be randomized and allocated into two intervention groups based on inclusion and exclusion criteria.Patients in group A will receive modified Otago exercises with conventional treatment.Patients in group B will receive Action Observation Training with conventional treatment.All participants will receive treatment of 40 minutes per session for 5 days a week for 8 weeks.The Michigan neuropathy screening instrument will be used for the assessment of diabetic neuropathy score.The strength,functional mobility and fall risk will be assessed by using 30 second chair stand test, Timed up and go test and fall efficacy scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes already diagnosed by physician from last 2 years
* Able to take instructions

Exclusion Criteria:

* Additional neurological problem Guillain barre syndrome, Parkinson disease, multiple sclerosis, other than neuropathy
* Participant with visual, vestibular system and auditory problems
* Participant with cardiovascular problem, cerebrovascular problem and epilepsy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Michigan neuropathy screening instrument (MNSI) | 6 months
  To determine neuropathy, Michigan neuropathy screening instrument (MNSI) developed by the researchers at the university of Michigan in 2000, used to diagnosed peripheral neuropathy. It includes two parts; section A is self-administered by the patient and assess the clinical symptoms through 15 Yes or No questions and section B is used on a clinical evaluation. The questionnaire inquiries about positive (pain, temperature sensation and tingling) and negative (numbness, sensory symptoms, cramps and muscle weakness, foot ulcer or cracks and amputation. Neuropathy can be defined as seven or more positive responses on the MNSI questionnaire. The test-retest reliability of the Turkish version of the MNSI was determined as 0.99 for the total score (intraclass correlation coefficient = 0.996)
30 second chair stand test | 6 months
  30 second chair stand test assesses the leg strength and endurance in older adults.it is part of the stop elderly accidents, deaths, and injuries which was created by centers for Disease Control and Preventions a screening tool for senior belonging to the high fall risk group .it has excellent test-retest reliability r=0.89(95%confident interval 0.79-0.93)The test measures the number of times and older adults can get up from a chair with their arms crossed in front of their trunk(on the opposite shoulder crossed at the wrists)in 30 seconds.
The timed up and go test | 6 months
  The timed up and go test is to identify mobility and balance. Patients sitting in a chair without armrest will be asked to stand up with the start command and walk the 3-meter distance, whose start and end points are specified before, turn around and sit on the chair again. The test will be repeated 3 times and the average time will be recorded. The TUG test showed excellent reliability (ICC>.95) The Timed -up and go‖ test showed good intrarater and interrater reliability (r = .93 ). less time taken by patient will be graded as good mobility
Fall Efficacy Scale International: | 6 months
  Fall Efficacy Scale International:
  It is a common test battery with 16 items that reveals the possibility of falling in patients. The total score ranges from 16 to 64, where 16 indicates NO concern and 64 indicates EXTREMELY concerned about falling during the performance of specific activities suggested by the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira JP, Sartor CD, Leal AM, Sacco IC, Sato TO, Ribeiro IL, Soares AS, Cunha JE, Salvini TF. The effect of peripheral neuropathy on lower limb muscle strength in diabetic individuals. Clin Biomech (Bristol). 2017 Mar;43:67-73. doi: 10.1016/j.clinbiomech.2017.02.003. Epub 2017 Feb 9. PMID 28213167
- [Background] Vratna E, Husakova J, Jarosikova R, Dubsky M, Woskova V, Bem R, Jirkovska A, Kralova K, Pyskova B, Lanska V, Fejfarova V. Effects of a 12-Week Interventional Exercise Programme on Muscle Strength, Mobility and Fitness in Patients With Diabetic Foot in Remission: Results From BIONEDIAN Randomised Controlled Trial. Front Endocrinol (Lausanne). 2022 Jul 5;13:869128. doi: 10.3389/fendo.2022.869128. eCollection 2022. PMID 35865313
- [Background] Van Eetvelde BLM, Lapauw B, Proot P, Vanden Wyngaert K, Celie B, Cambier D, Calders P. The impact of sensory and/or sensorimotor neuropathy on lower limb muscle endurance, explosive and maximal muscle strength in patients with type 2 diabetes mellitus. J Diabetes Complications. 2020 Jun;34(6):107562. doi: 10.1016/j.jdiacomp.2020.107562. Epub 2020 Feb 24. PMID 32122790